CLINICAL TRIAL: NCT00790400
Title: A Randomized, Double-blind, Placebo-controlled Study of RAD0001 in the Treatment of Angiomyolipoma in Patients With Either Tuberous Sclerosis Complex (TSC) or Sporadic Lymphangioleiomyomatosis (LAM)
Brief Title: Efficacy and Safety of RAD001 in Patients Aged 18 and Over With Angiomyolipoma Associated With Either Tuberous Sclerosis Complex (TSC) or Sporadic Lymphangioleiomyomatosis (LAM)
Acronym: EXIST-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRAD001M2302; 2008-002113-48 (EudraCT Number)
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-01

CONDITIONS: Tuberous Sclerosis Complex (TSC); Lymphangioleiomyomatosis (LAM)
Keywords: Angiomyolipoma; AML; Tuberous Sclerosis Complex; TSC; mTOR; RAD001; Mammalian Target of Rapamycin; Everolimus; Afinitor; SEGA; Subependymal Giant Cell Astrocytoma; Seizures; Tuberous sclerosis complex (TSC); Tuberous sclerosis; benign tumors of brain; kidney; heart; eyes; lungs; skinTSC1; TSC2; hamaratin; tuberin, tumor growth suppressors; gyri; tubers; Sporadic Lymphangioleiomyomatosis.; Lymphangioleiomyomatosis (LAM); rare lung disease
MeSH Terms: conditions — Tuberous Sclerosis; Lymphangioleiomyomatosis; Angiomyolipoma; Hereditary Sensory and Autonomic Neuropathies; Astrocytoma; Seizures; Tuberous Sclerosis 2 | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus (Experimental): Study drug was given by continuous oral daily dosing of two 5 mg tablets.
  Interventions: Drug: Everolimus (RAD001)
- Placebo (Placebo Comparator): Placebo was given by continuous oral daily dosing of two 5 mg tablets.
  Interventions: Drug: Everolimus Placebo

INTERVENTIONS:
Drug: Everolimus (RAD001) — Everolimus is used in 5 mg strength tablets, blister-packed under aluminum foil in units of ten tablets and dosed on a daily basis. 10mg daily dosing throughout the trial.
  Other Names: RAD001
  Arms: Everolimus
Drug: Everolimus Placebo — Matching placebo was provided as a matching tablet and was also blister-packed under aluminum foil in units of ten.
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of RAD001 in treating patients with Angiomyolipoma associated with Tuberous Sclerosis Complex or Sporadic Lymphangioleiomyomatosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18 years or older
* Clinically definite diagnosis of Tuberous Sclerosis Complex according to the modified Gomez criteria or sporadic LAM (biopsy-proven or compatible chest CT scan)
* Clinically definite diagnosis of renal angiomyolipoma
* At least one Angiomyolipoma of ≥ 3 cm in its longest diameter using CT or MRI
* Females of child bearing potential must use birth control and have documentation of negative pregnancy test
* Written informed consent according to local guidelines

Exclusion Criteria:

* Recent heart attack, cardiac related chest pain or stroke
* Severely impaired lung function
* Bleeding related to angiomyolipoma or embolization during 6 months prior to randomization
* Clinically significant chylous ascites
* Clinically significant hematological or hepatic abnormality
* Severe liver dysfunction
* Severe kidney dysfunction
* Pregnancy or breast feeding
* Current infection
* History of organ transplant
* Surgery within two months prior to study enrollment
* Prior therapy with a medication in the same class as Everolimus
* Recent use of an investigational drug
* Bleeding diathesis or on oral anti-vitamin K medication
* Uncontrolled high cholesterol
* Uncontrolled diabetes
* HIV
* Inability to attend scheduled clinic visits
* Patients with metal implants thus prohibiting MRI evaluations
* Angiomyolipoma which requires surgery at the time of randomization
* History of malignancy
* Severe or uncontrolled medical conditions which would cause an unacceptable safety risk or compromise compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Tuberous Sclerosis Center, Phoenix, Arizona
  - Massachusetts General Hospital Massachussetts General Hospita, Boston, Massachusetts
  - Minnesota Epilepsy Group, Saint Paul, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - LeBonheur Childrens Medical Group SC-2, Memphis, Tennessee
- Novartis Investigative Site, Torono, Ontario, Canada
- Novartis Investigative Site, Lyon, France, France
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, München
- Italy (3):
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Roma
- Japan (3):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Yamagata, Yamagata
- Novartis Investigative Site, Utrecht, Netherlands, Netherlands
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- United Kingdom (4):
  - Novartis Investigative Site, Brighton, East Sussex
  - Novartis Investigative Site, Craigavon, Northern Ireland
  - Novartis Investigative Site, Cardiff, Wales
  - Novartis Investigative Site, London

REFERENCES:
- [Background] Bissler JJ, Kingswood JC, Radzikowska E, Zonnenberg BA, Frost M, Belousova E, Sauter M, Nonomura N, Brakemeier S, de Vries PJ, Whittemore VH, Chen D, Sahmoud T, Shah G, Lincy J, Lebwohl D, Budde K. Everolimus for angiomyolipoma associated with tuberous sclerosis complex or sporadic lymphangioleiomyomatosis (EXIST-2): a multicentre, randomised, double-blind, placebo-controlled trial. Lancet. 2013 Mar 9;381(9869):817-24. doi: 10.1016/S0140-6736(12)61767-X. PMID 23312829
- [Derived] Bissler JJ, Nonomura N, Budde K, Zonnenberg BA, Fischereder M, Voi M, Louveau AL, Herbst F, Bebin EM, Curatolo P, Zonta A, Belousova E. Angiomyolipoma rebound tumor growth after discontinuation of everolimus in patients with tuberous sclerosis complex or sporadic lymphangioleiomyomatosis. PLoS One. 2018 Sep 7;13(9):e0201005. doi: 10.1371/journal.pone.0201005. eCollection 2018. PMID 30192751
- [Derived] Bissler JJ, Budde K, Sauter M, Franz DN, Zonnenberg BA, Frost MD, Belousova E, Berkowitz N, Ridolfi A, Christopher Kingswood J. Effect of everolimus on renal function in patients with tuberous sclerosis complex: evidence from EXIST-1 and EXIST-2. Nephrol Dial Transplant. 2019 Jun 1;34(6):1000-1008. doi: 10.1093/ndt/gfy132. PMID 30053159
- [Derived] Sparagana S, Franz DN, Krueger DA, Bissler JJ, Berkowitz N, Burock K, Kingswood JC. Pooled analysis of menstrual irregularities from three major clinical studies evaluating everolimus for the treatment of tuberous sclerosis complex. PLoS One. 2017 Oct 12;12(10):e0186235. doi: 10.1371/journal.pone.0186235. eCollection 2017. PMID 29023494
- [Derived] Bissler JJ, Kingswood JC, Radzikowska E, Zonnenberg BA, Frost M, Belousova E, Sauter M, Nonomura N, Brakemeier S, de Vries PJ, Berkowitz N, Miao S, Segal S, Peyrard S, Budde K. Everolimus for renal angiomyolipoma in patients with tuberous sclerosis complex or sporadic lymphangioleiomyomatosis: extension of a randomized controlled trial. Nephrol Dial Transplant. 2016 Jan;31(1):111-9. doi: 10.1093/ndt/gfv249. Epub 2015 Jul 8. PMID 26156073
- See also: Visit EXIST-2 NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/webapp/portals/EXISTClinicalTrials/page.do

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multicenter trial conducted at 24 sites in 11 countries. As the primary analysis of the core phase of the study favored everolimus over placebo, an open-label extension phase started: patients randomized in placebo were offered to switch on everolimus and those still receiving everolimus at the end of the core phase could continue the treatment.
Pre-assignment Details: The trial had a 2:1 randomization in favor of the everolimus arm. 118 patients were randomized to the core phase of the study. 112 patients received everolimus during core and/or extension phase.
Period: Double-blind Period (Core Phase)
Arm/Group | Everolimus | Placebo
Started | 79 | 39
Completed | 72 (Completed = Completed the Core phase & moved to Extension phase) | 26 (Completed = 1st received Placebo in the Core phase, switched to Everolimus in Extension phase)
Not Completed | 7 | 13
Not completed — Protocol Violation | 1 | 0
Not completed — Progressive disease | 0 | 9
Not completed — Adverse Event | 2 | 4
Not completed — Abnormal lab value (s) | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Administrative problems | 1 | 0
Not completed — Death | 1 | 0
Period: Everolimus Period (Core or Extension)
Arm/Group | Everolimus | Placebo
Started | 112 (112 pts had Everolimus during core and/or extension (6 from placebo did not switch to Eve. in ext.)) | 0 (Placebo randomized patients who switched to Everolimus are reported in "Everolimus" arm.)
Completed | 83 (Treatment duration completed as per protocol) | 0
Not Completed | 29 | 0
Not completed — Adverse Event | 9 | 0
Not completed — Abnormal lab value (s) | 1 | 0
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Administrative problems | 2 | 0
Not completed — Death | 1 | 0
Not completed — Disease progression | 5 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — New treatment | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus | Placebo | Total
Number analyzed (Participants) | 79 | 39 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (10.37) | 31.0 (9.64) | 32.0 (10.12)
Age, Customized [Number; unit: Participants]
  <30 years | 35 | 20 | 55
  ≥ 30 years | 44 | 19 | 63
Gender [Count of Participants; unit: Participants]
  Female | 52 | 26 | 78
  Male | 27 | 13 | 40

OUTCOME MEASURES:

1. Primary Outcome: Angiomyolipoma Response Rate as Per Central Radiology Review
Description: Angiomyolipoma response defined as the combination of the following criteria: reduction in angiomyolipoma volume of ≥ 50% relative to baseline, where angiomyolipoma volume was sum of volumes of all target lesions identified at baseline, and with a confirmatory scan performed approximately 12 weeks later (no sooner than 8 weeks later); no new angiomyolipoma lesions ≥ 1.0 cm in longest diameter were identified; there were no kidney increases in volume > 20% from nadir. The patient did not have any angiomyolipoma-related bleeding of ≥ grade 2.
  For the everolimus (core/extension periods) treatment group, the baseline means the latest value on or before starting everolimus.
Time Frame: From date of randomization until the earliest date of first documented AML progression, date of further anti-AML medication (including open-label Everolimus)/surgery or up to 5.7 years
Population: The Full Analysis Set (FAS) is defined according to the Intention-to-Treat principle and consists of all randomized patients.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Everolimus Randomized (Core Period): Study drug was given by continuous oral daily dosing of two 5 mg tablets.
- Placebo Randomized (Core Period): Placebo was given by continuous oral daily dosing of two 5 mg tablets.
- Everolimus (Core and/or Extension Period): Patients initially randomized in everolimus and patients initially randomized in placebo but who crossed-over to everolimus during extension.
Arm/Group | Everolimus Randomized (Core Period) | Placebo Randomized (Core Period) | Everolimus (Core and/or Extension Period)
Number analyzed (Participants) | 79 | 39 | 112
Percentage of Participants | 41.8 [30.8 to 53.4] | 0 [0.0 to 9.0] | 58.0 [48.3 to 67.3]
Statistical Analysis 1: Comparison: Everolimus Randomized (Core Period) vs Placebo Randomized (Core Period); Test type: Superiority or Other; p < 0.0001, Clopper-Pearson

2. Secondary Outcome: Time to Angiomyolipoma Progression as Per Central Radiology Review
Description: Time to angiomyolipoma progression (TTAP) is defined as time from date of randomization to date of first documented angiomyolipoma progression. Angiomyolipoma progression was defined as one or more of the following: Increase from nadir of ≥ 25% in angiomyolipoma volume to value greater than baseline; the appearance of a new angiomyolipoma ≥ 1.0 cm in longest diameter; an increase from nadir of 20% or more in the volume of either kidney to a value greater than baseline; angiomyolipoma-related bleeding grade ≥ 2.
  For the everolimus (core/extension periods) treatment group, the time to angiomyolipoma progression is defined starting from the start of everolimus. The baseline means the latest value on or before starting everolimus.
Time Frame: From date of randomization until the earliest date of first documented AML progression, date of further anti-AML medication (including open-label Everolimus)/surgery or up to about 5.7 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus Randomized (Core Period) | Placebo Randomized (Core Period) | Everolimus (Core and/or Extension Period)
Number analyzed (Participants) | 79 | 39 | 112
months | NA [NA to NA] — Median not reached since too few number of patients with progressions (n=3). | 11.37 [11.07 to NA] — Upper limit not estimable due to few number of patients at this time point. | NA [NA to NA] — Median not reached since too few number of patients with progressions (n=16)

3. Secondary Outcome: Skin Lesion Response Rate as Per Investigator (Only Patients With at Least One Skin Lesion at Baseline)
Description: Skin lesion response rate in the double-blind period was determined only among patients with at least one skin lesion at baseline, and is the percentage of this group of patients with a best overall skin lesion response on the Physician's Global Assessment of Clinical Condition (PGA) of either complete clinical response (CCR) or partial response (PR). A complete clinical response (CCR) requires a grading of 0 indicating the absence of disease (histological confirmation is not required). Grades 1, 2, and 3 constitute partial response, indicating improvement of at least 50 percent, but less than 100 percent improvement. For the everolimus (core/extension periods) treatment group, the baseline means the latest value on or before starting everolimus.
Time Frame: as for outcome 1
Population: The Full Analysis Set (FAS) is defined according to the Intention-to-Treat principle and consists of all randomized patients. Only patients with at least one skin lesion at baseline are included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus Randomized (Core Period) | Placebo Randomized (Core Period) | Everolimus (Core and/or Extension Period)
Number analyzed (Participants) | 77 | 37 | 112
Percentage of participants | 26 [16.6 to 37.2] | 0 [0.0 to 9.5] | 68.2 [58.5 to 76.9]

4. Secondary Outcome: Percentage of Participants With Renal Impairment
Description: Renal Impairment was measured by glomerular filtration rate which was calculated using the Modification of Diet in Renal Disease formula. Percentage of participants with renal impairment was reported. Severe renal impairment was defined as a GFR of <30ml/min/1.73m2.
Time Frame: Day 1 up to 28 days after end of treatment
Population: Safety set consists of all patients who received at least 1 dose of the double-blind study drug with a valid post-baseline assessment. For the everolimus (core/extension) treatment arm, patients received at least 1 dose of everolimus with a valid post-baseline assessment, where baseline was defined as the assessment just before start of everolimus.
Measure: Number; unit: Percentage of Participants
Arm/Group | Everolimus Randomized (Core Period) | Placebo Randomized (Core Period) | Everolimus (Core and/or Extension Period)
Number analyzed (Participants) | 79 | 39 | 112
Percentage of Participants
  Glomerular filtration rate <30 ml/min/1.73m^2 | 2.5 | 7.7 | 7.1
  Glomerular filtration rate≥ 30 ml/min/1.73m^2 | 97.5 | 92.3 | 92.9

5. Secondary Outcome: Change From Baseline in Plasma Angiogenic Molecules - Vascular Endothelial Growth Factor (VEGF) Marker
Description: Blood samples for biomarker assessment were collected immediately prior to study administration. On-treatment samples was compared to baseline samples with the change from baseline.
Time Frame: 4 weeks, 12 weeks, 24 weeks, 36 weeks 48 weeks, 60 weeks, 72 weeks
Population: The Full Analysis Set (FAS) is defined according to the Intention-to-Treat principle and consists of all randomized patients. The 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Everolimus Randomized (Core Period) | Placebo Randomized (Core Period)
Number analyzed (Participants) | 79 | 39
pg/mL
  Week 4 (n:56, 28) | 38.7 (141.89) | 17.6 (57.51)
  Week 12 (n:56, 29) | 43.4 (60.62) | -6.1 (46.28)
  Week 24 (n:53, 29) | 31.1 (75.83) | -4.3 (44.76)
  Week 36 (n:26, 18) | 18.0 (45.07) | 5.4 (24.01)
  Week 48 (n:16, 8) | 55.3 (80.31) | 3.1 (34.55)
  Week 60 (n:0, 1) | NA (NA) — N/A = No patient was included at this time point, so no mean, no standard deviation (SD) could be calculated. | -4.12 (NA) — N/A = only 1 patient was included, so no SD could be calculated
  Week 72 (n:0, 1) | NA (NA) — N/A = No patient was included at this time point, so no mean, no SD could be calculated. | -6.1 (NA) — N/A = only 1 patient was included, so no SD could be calculated

6. Secondary Outcome: Everolimus Trough Concentrations (Cmin)
Description: Cmin values collected prior to dose administration on the same study day and at 20-28 hours after previous dose, at steady state, and patient did not vomit within 4 hours of previous dose. Samples collected during the first 4 days of dosing were excluded from all analyses.
Time Frame: Prior to dosing at weeks 2, 4, 12, 24, 48
Population: The analysis was performed in the Safety Set population for patients treated only with Everolimus and with a confirmed PK sample.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Everolimus Randomized (Core Period)
Number analyzed (Participants) | 79
ng/mL
  Prior to dosing at Week 2 (n:43) | 7.63 (4.32)
  Prior to dosing Week 4 (n:44) | 7.72 (4.35)
  Prior to dosing Week 12 (n:49) | 8.79 (6.75)
  Prior to dosing Week 24 (n:46) | 9.37 (8.83)
  Prior to dosing Week 48 (n:15) | 11.49 (12.01)

7. Secondary Outcome: Everolimus Blood Concentrations (C2h) at 2 Hours Post-dose
Description: C2h values collected 1-3 hours after dose administration on the same study day, at steady state, and patient did not vomit between taking previous dose and blood collection. Samples collected during the first 4 days of dosing will be excluded from all analyses.
Time Frame: 2 hours post-dose administration at Weeks 2, 4, 12, 24, 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Everolimus Randomized (Core Period)
Number analyzed (Participants) | 79
ng/mL
  2 hours post dose administration at Week 2 (n:55) | 33.38 (15.66)
  2 hours post dose administration at Week 4 (n:49) | 30.89 (14.96)
  2 hours post dose administration at Week 12 (n:56) | 34.48 (15.10)
  2 hours post dose administration at Week 24 (n:50) | 39.27 (22.25)
  2 hours post dose administration at Week 48 (n:14) | 33.20 (18.45)

8. Secondary Outcome: Time to Angiomyolipoma Response - Only Everolimus Patients With Angiomyolipoma Response
Description: Time to angiomyolipoma response was defined as the time from the date of randomization until the date of the first documented angiomyolipoma response. Angiomyolipoma response defined as the combination of the following criteria: reduction in angiomyolipoma volume of ≥ 50% relative to baseline, where angiomyolipoma volume was sum of volumes of all target lesions identified at baseline, and with a confirmatory scan performed approximately 12 weeks later (no sooner than 8 weeks later); no new angiomyolipoma lesions ≥ 1.0 cm in longest diameter were identified; no kidney increases in volume > 20% from nadir; no angiomyolipoma-related bleeding of ≥ grade 2.
  For the everolimus (core/extension periods) treatment group, the time to angiomyolipoma response is from the start of everolimus. The baseline in the response definition means the latest value on or before starting everolimus.
Time Frame: as for outcome 1
Population: The analysis was performed on the Full analysis Set for patients in Everolimus arm and who experienced an angiomyolipoma response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus Randomized (Core Period) | Everolimus (Core and/or Extension Period)
Number analyzed (Participants) | 33 | 65
months | 2.86 [2.79 to 3.02] | 2.89 [2.79 to 3.19]

9. Secondary Outcome: Duration of Angiomyolipoma Response - Only Everolimus Patients With Angiomyolipoma Response
Description: Duration of angiomyolipoma response was defined as the time from the date of the first documented angiomyolipoma response until the date of the first documented angiomyolipoma progression . Angiomyolipoma response was defined as the combination of the following criteria: reduction in angiomyolipoma volume of ≥ 50% relative to baseline, where angiomyolipoma volume was sum of volumes of all target lesions identified at baseline, and with a confirmatory scan performed approximately 12 weeks later (no sooner than 8 weeks later); no new angiomyolipoma lesions ≥ 1.0 cm in longest diameter were identified; there were no kidney increases in volume > 20% from nadir. The patient did not have any angiomyolipoma-related bleeding of ≥ grade 2.
Time Frame: as for outcome 2
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus Randomized (Core Period) | Everolimus (Core and/or Extension Period)
Number analyzed (Participants) | 33 | 65
months | NA [NA to NA] — N/A = Median not reached since no patients progressed | NA [NA to NA] — N/A = Median not reached since too few no of patients with progressions (n=2)

10. Secondary Outcome: Duration of Skin Lesion Response - Only Everolimus Patients With Best Overall Skin Lesion Response of Complete Clinical Response (CCR) or Partial Response (PR)
Description: Duration of skin lesion response is defined as the time from the date of the first skin lesion response until the date of the first skin lesion progression, according to the PGA (physician's global assessment of clinical condition). A progression is when the disease is worse than at baseline evaluation by >=25% or more.
Time Frame: as for outcome 2
Population: The analysis was performed on the Full analysis Set for patients in Everolimus arm and who experienced a best overall skin lesion response CCR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus Randomized (Core Period) | Everolimus (Core and/or Extension Period)
Number analyzed (Participants) | 20 | 73
months | NA [NA to NA] — N/A = Median not reached since no patients progressed | NA [NA to NA] — N/A = Median not reached since no patients progressed

ADVERSE EVENTS:
Groups:
- Everolimus Randomized (Core & Ext): Patients who were randomized and treated with Everolimus during the Core and Extension phase
- Placebo Randomized/Crossed Over to Everolimus: Patients who were randomized to placebo in the Core phase and who crossed-over to Everolimus in the Extension phase
- Placebo Randomized/Never Crossed-over: Patients randomized to placebo who never crossed-over to Everolimus
Arm/Group | Everolimus Randomized (Core & Ext) | Placebo Randomized/Crossed Over to Everolimus | Placebo Randomized/Never Crossed-over
Serious Adverse Events (participants affected / at risk) | 28/79 | 17/33 | 3/6
Other Adverse Events (participants affected / at risk) | 79/79 | 33/33 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus Randomized (Core & Ext) (N=79) | Placebo Randomized/Crossed Over to Everolimus (N=33) | Placebo Randomized/Never Crossed-over (N=6)
Bone marrow oedema (Blood and lymphatic system disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Incision site infection (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Complex regional pain syndrome (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Diplegia (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 3 | 3 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 2 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 1
Psychiatric decompensation (Psychiatric disorders) | 0 | 1 | 0
Psychogenic seizure (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0
Renal haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Breast hypoplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Haemodynamic instability (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus Randomized (Core & Ext) (N=79) | Placebo Randomized/Crossed Over to Everolimus (N=33) | Placebo Randomized/Never Crossed-over (N=6)
Anaemia (Blood and lymphatic system disorders) | 9 | 6 | 0
Leukopenia (Blood and lymphatic system disorders) | 9 | 7 | 0
Lymphopenia (Blood and lymphatic system disorders) | 5 | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 7 | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 3 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 2 | 0
Hamartoma (Congenital, familial and genetic disorders) | 1 | 3 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 13 | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 7 | 4 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 19 | 12 | 1
Constipation (Gastrointestinal disorders) | 8 | 6 | 1
Dental caries (Gastrointestinal disorders) | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 17 | 11 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 0 | 0
Flatulence (Gastrointestinal disorders) | 5 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 15 | 4 | 1
Nausea (Gastrointestinal disorders) | 18 | 7 | 2
Stomatitis (Gastrointestinal disorders) | 41 | 10 | 0
Toothache (Gastrointestinal disorders) | 5 | 3 | 0
Vomiting (Gastrointestinal disorders) | 18 | 5 | 0
Asthenia (General disorders) | 2 | 2 | 0
Fatigue (General disorders) | 17 | 13 | 1
Influenza like illness (General disorders) | 2 | 5 | 1
Malaise (General disorders) | 0 | 2 | 0
Oedema peripheral (General disorders) | 16 | 10 | 0
Pyrexia (General disorders) | 11 | 6 | 1
Hypersensitivity (Immune system disorders) | 1 | 2 | 0
Seasonal allergy (Immune system disorders) | 3 | 2 | 0
Bronchitis (Infections and infestations) | 9 | 9 | 1
Cellulitis (Infections and infestations) | 2 | 4 | 0
Conjunctivitis (Infections and infestations) | 4 | 2 | 0
Ear infection (Infections and infestations) | 5 | 1 | 0
Folliculitis (Infections and infestations) | 4 | 1 | 0
Furuncle (Infections and infestations) | 4 | 2 | 0
Gastroenteritis (Infections and infestations) | 9 | 4 | 0
Gastroenteritis viral (Infections and infestations) | 4 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 2 | 0
Gingivitis (Infections and infestations) | 2 | 3 | 0
Influenza (Infections and infestations) | 8 | 3 | 1
Nasopharyngitis (Infections and infestations) | 36 | 19 | 1
Oral candidiasis (Infections and infestations) | 1 | 2 | 0
Oral herpes (Infections and infestations) | 5 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 3 | 0
Otitis media (Infections and infestations) | 6 | 2 | 0
Periodontitis (Infections and infestations) | 6 | 0 | 0
Pharyngitis (Infections and infestations) | 5 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 5 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 2 | 0
Rash pustular (Infections and infestations) | 7 | 3 | 0
Respiratory tract infection (Infections and infestations) | 5 | 2 | 0
Respiratory tract infection viral (Infections and infestations) | 5 | 0 | 0
Rhinitis (Infections and infestations) | 7 | 6 | 1
Sinusitis (Infections and infestations) | 11 | 4 | 1
Tonsillitis (Infections and infestations) | 1 | 6 | 0
Tooth abscess (Infections and infestations) | 7 | 2 | 0
Tooth infection (Infections and infestations) | 4 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 15 | 4 | 0
Urinary tract infection (Infections and infestations) | 25 | 12 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 3 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 2 | 1
Activated partial thromboplastin time prolonged (Investigations) | 10 | 5 | 0
Alanine aminotransferase increased (Investigations) | 9 | 5 | 0
Aspartate aminotransferase increased (Investigations) | 10 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 11 | 5 | 0
Blood cholesterol increased (Investigations) | 11 | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 5 | 0
Blood creatinine increased (Investigations) | 4 | 4 | 0
Blood fibrinogen increased (Investigations) | 4 | 5 | 0
Blood lactate dehydrogenase increased (Investigations) | 9 | 4 | 0
Blood phosphorus decreased (Investigations) | 6 | 1 | 0
Blood triglycerides increased (Investigations) | 10 | 4 | 0
C-reactive protein increased (Investigations) | 3 | 2 | 0
Carbon monoxide diffusing capacity decreased (Investigations) | 7 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 5 | 1 | 0
Haemoglobin decreased (Investigations) | 11 | 3 | 0
International normalised ratio increased (Investigations) | 4 | 3 | 0
Low density lipoprotein increased (Investigations) | 1 | 2 | 0
Weight decreased (Investigations) | 7 | 4 | 0
Weight increased (Investigations) | 4 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 6 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 29 | 11 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 10 | 5 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 8 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 5 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 15 | 4 | 0
Iron deficiency (Metabolism and nutrition disorders) | 7 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 14 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 7 | 0
Convulsion (Nervous system disorders) | 8 | 4 | 0
Dizziness (Nervous system disorders) | 9 | 4 | 1
Epilepsy (Nervous system disorders) | 3 | 2 | 0
Headache (Nervous system disorders) | 26 | 15 | 0
Lethargy (Nervous system disorders) | 1 | 2 | 0
Migraine (Nervous system disorders) | 9 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 0
Petit mal epilepsy (Nervous system disorders) | 4 | 2 | 0
Affective disorder (Psychiatric disorders) | 0 | 2 | 0
Aggression (Psychiatric disorders) | 1 | 3 | 0
Anxiety (Psychiatric disorders) | 4 | 1 | 0
Depression (Psychiatric disorders) | 8 | 4 | 0
Insomnia (Psychiatric disorders) | 6 | 1 | 0
Mood swings (Psychiatric disorders) | 3 | 2 | 0
Sleep disorder (Psychiatric disorders) | 2 | 3 | 0
Haematuria (Renal and urinary disorders) | 2 | 3 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 11 | 10 | 0
Renal pain (Renal and urinary disorders) | 0 | 2 | 0
Amenorrhoea (Reproductive system and breast disorders) | 16 | 6 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 11 | 2 | 0
Menstruation irregular (Reproductive system and breast disorders) | 11 | 4 | 0
Metrorrhagia (Reproductive system and breast disorders) | 4 | 3 | 0
Ovarian cyst (Reproductive system and breast disorders) | 5 | 3 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 7 | 5 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 7 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 3 | 0
Lymphangioleiomyomatosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 6 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 25 | 11 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 5 | 0
Eczema (Skin and subcutaneous tissue disorders) | 11 | 3 | 0
Papule (Skin and subcutaneous tissue disorders) | 4 | 2 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 4 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 3 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Circulatory collapse (Vascular disorders) | 2 | 2 | 0
Haematoma (Vascular disorders) | 2 | 2 | 0
Hypertension (Vascular disorders) | 22 | 12 | 0
Lymphoedema (Vascular disorders) | 4 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.